CLINICAL TRIAL: NCT07405294
Title: A Retrospective Cohort Study Comparing Clinical Outcomes and Unscheduled Follow-up of Telemedicine and In-person Medication Abortion
Brief Title: TeleMAb Retrospective Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Erika Levi, MD, Wyeth-Ayerst Associate Professor of Women's Health in Obstetrics and Gynecology, Columbia University
Other Study IDs: AAAV5073
Record Dates: First submitted 2026-02-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Medication Abortion; Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Telemedicine Med Ab: Patients who received medication abortion through the telemedicine medication abortion service during the study period.
  Interventions: Other: Telemedicine Medication Abortion
- In-person Med Ab: Patients who received an in-person medication abortion at the clinic during the study period.

INTERVENTIONS:
Other: Telemedicine Medication Abortion — Meeting with a clinician via video visit to determine if patient is eligible for medication abortion without pre-treatment ultrasound or laboratory testing. If eligible, the patient travels to clinic to pick up medications in person.
  Groups: Telemedicine Med Ab

SUMMARY:
The objective of this study is to evaluate whether there are different clinical outcomes and unscheduled follow-ups between in-person and telemedicine medication abortion, and to better understand patients' experiences with telemedicine medication abortion and their motivations for seeking unscheduled follow-up care in a setting where abortion care, including both virtual and in-person follow-up care, is readily accessible.

DETAILED DESCRIPTION:
This study will be retrospective chart review comparing clinical and demographic characteristics, eligibility, treatment success, participation in unscheduled and scheduled follow-ups, and adverse events of patients who obtained a telemedicine medication abortion through the Telehealth Medication Abortion Clinic with patients who received an in-person medication abortion provided at the Family Planning Faculty Practice from June 2023 through September 2024.

ELIGIBILITY:
Inclusion Criteria:

* Received telemedicine or in-person medication abortion at Columbia University Irving Medical Center's associated practices from June 12, 2023 through September 30, 2024
* Gestational age <70 days (based on best obstetrical dating)
* English or Spanish speaking

Exclusion Criteria:

* Received mifepristone and misoprostol for early pregnancy loss
* Patient determined to have contraindication to medication abortion
* Opted for procedural management instead of medication abortion
* Decided to continue with the pregnancy
* Presenting for a second medication abortion at CUIMC during the study period
* Non-English or Spanish speaking

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Biologically female patients of reproductive age with an unwanted pregnancy seeking care at Columbia University's family planning clinics and interested in medication abortion.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of unscheduled follow-ups | 3 months after initial encounter
  If patients engaged in follow-up are outside of their routinely scheduled follow-up visit 1-2 weeks after medication abortion

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No